CLINICAL TRIAL: NCT06451666
Title: A Phase 3, Multicenter, Double-Masked, Randomized, Vehicle-Controlled Study Evaluating the Safety and Efficacy of Pilocarpine HCl in Participants With Presbyopia
Brief Title: Safety and Efficacy Study of Pilocarpine HCl Ophthalmic Solution in Participants With Presbyopia
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: CSPC Ouyi Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SYH9042-001
Record Dates: First submitted 2024-05-29; First posted 2024-06-11 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-05

CONDITIONS: Presbyopia
MeSH Terms: conditions — Presbyopia

STUDY DESIGN:
Intervention Model Description: For arm 1, patients received pilocarpine HCl ophthalmic solution 1.25%, one drop in each eye, once daily, for up to 30 days.
  For arm 2, patients received vehicle, one drop in each eye, once daily, for up to 30 days.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Pilocarpine HCl Ophthalmic Solution (Experimental)
  Interventions: Drug: Pilocarpine HCl Ophthalmic Solution
- Vehicle (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Pilocarpine HCl Ophthalmic Solution — Pilocarpine HCl ophthalmic solution 1.25%, one drop in each eye, once daily, for up to 30 days
  Arms: Pilocarpine HCl Ophthalmic Solution
Drug: Vehicle — Vehicle, one drop in each eye, once daily, for up to 30 days.
  Arms: Vehicle

SUMMARY:
A study to evaluate the efficacy, safety, and pharmacokinetics of pilocarpine HCl ophthalmic solution when administered bilaterally, once daily for 30 days in participants with presbyopia.

ELIGIBILITY:
Inclusion Criteria:

* 1 Participant must be 40 to 65 years of age inclusive, at the time of the screening visit;
* 2 Emmetropes or non-emmetropes with best distance correction in the range of spherical -4.00 D to +2.00 D inclusively and cylinder ±2.00 D with photopic, high contrast CDVA of 20/25 or better in each eye at the screening and baseline visits;
* 3 Mesopic, high contrast DCNVA of 20/40 to 20/100 in each eye at the screening and baseline visits;
* 4 Photopic, high contrast, near visual acuity correctable to 20/40 or better in each eye at the screening and baseline visits;
* 5 Dark adaptation pupil diameter between 4.0 mm and 8.0 mm in both eyes at the screening visit;
* 6 Capable of giving signed informed consent, which includes compliance with the requirements and restrictions listed in the ICF and in this protocol.

Exclusion Criteria:

* 1 Clinically significant disease state, in the opinion of the examining investigator or designee, in any body system;
* 2 Known allergy or sensitivity to the study intervention or its components or other cholinergic agonist medications;
* 3 Any active ocular inflammation within 30 days prior to the first use of the investigational drug;
* 4 Current enrollment in an study or participation in such a study within 30 days prior to the first use of the investigational drug;
* 5 Any clinical condition or previous surgery that might affect the absorption, distribution, biotransformation, or excretion;
* 6 History of cataract surgery, phakic intraocular lens surgery, corneal refractive surgery, radial keratotomy, or any intraocular surgery;
* 7 Presence of any ocular condition that, in the opinion of the investigator, could affect the safety of the participant or interpretation of efficacy parameters;
* 8 Moderate to severe dry eye disease at the screening visit;
* 9 Lens opacity in either eye that is determined to cause significant disturbance of the central visual axis at the screening visit;
* 10 Diagnosis of any type of glaucoma or ocular hypertension;
* 11 Female who have a positive pregnancy test during the screening period, lactating, or planning a pregnancy during the study.

Ages: 40 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 330 (Estimated)
Dates: Start 2024-06-30 (Estimated); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Title: Percentage of Participants Gaining 3 Lines or More in Mesopic, High-contrast, Binocular Distance-Corrected Near Visual Acuity (DCNVA) at Day 30, Hour 3 | Baseline (Day 1) to Day 30 (Hour 3)

SECONDARY OUTCOMES:
Incidence and frequency of adverse events (AE) and serious adverse events (SAE) etc. | Through study completion, an average of 60 days
Area under the plasma concentration time curve from time zero to the last measurable concentration(AUC0-t) | Day 1 and Day 30
Area under the plasma concentration-time curve from time zero to infinity(AUC0-inf) | Day 1 and Day 30
Maximum plasma concentration(Cmax) | Day 1 and Day 30
Time to maximum plasma concentration (Tmax) | Day 1 and Day 30
Apparent Volume of Distribution During Terminal Phase (Vz/F) | Day 1 and Day 30
Apparent Terminal Elimination Half-Life (T1/2) | Day 1 and Day 30
Apparent total body clearance (CL/F) | Day 1 and Day 30